CLINICAL TRIAL: NCT01934894
Title: Phase II Study With Lead-in Safety Cohort of Cabazitaxel Plus Lapatinib as Therapy for HER2-Positive Metastatic Breast Cancer Patients With Intracranial Metastases
Brief Title: Cabazitaxel Plus Lapatinib as Therapy for HER2-Positive Metastatic Breast Cancer Patients With Intracranial Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of significant signal of efficacy
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry); GlaxoSmithKline (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 200
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Metastatic Breast Cancer With Intracranial Metastases
Keywords: HER2-positive breast cancer; intracranial metastases; lapatinib; cabazitaxel
MeSH Terms: interventions — cabazitaxel; XRP6258; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cabazitaxel and lapatinib combination (Experimental): * Cabazitaxel 1-hour IV infusion on Day 1 of each 3 week cycle (dose to be determined)
  * Lapatinib PO once daily (dose to be determined)
  Treatment cycles will be repeated every 3 weeks.
  Interventions: Drug: cabazitaxel; Drug: lapatinib

INTERVENTIONS:
Drug: cabazitaxel
  Other Names: Jevtana; XRP6258
Drug: lapatinib
  Other Names: Tykerb; GW572016

SUMMARY:
This phase II trial will combine two agents, cabazitaxel and lapatinib, to treat patients with metastatic breast cancer (MBC) which has metastasized to the brain. The first portion of the study will determine the optimal dose of the cabazitaxel/lapatinib combination to administer to patients. After determining the optimal dose, patients will continue treatment with cabazitaxel and lapatinib to assess response to treatment with these agents.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, Phase II study with a lead-in safety cohort. Through the safety lead-in portion of this trial we will define the optimal dose of cabazitaxel when given in combination with lapatinib for patients with HER2-positive MBC and CNS metastases. The Phase II portion will further assess intracranial response rate in patients with HER2-positive MBC and CNS metastases. Toxicity and progression free survival (PFS) will be obtained and evaluated. The trial will be conducted at multiple study sites by SCRI Development Innovations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2-positive MBC and unequivocal evidence of brain metastases.
2. Documented HER2-positive tumor status at study entry defined as:

   * Immunohistochemical (IHC) score 3+ or
   * IHC score 1-2+ and confirmed as FISH (Fluorescence in situ hybridization) positive (based on ASCO-CAP guidelines 2013) or
   * FISH or ISH (in situ hybridization) positive (based on ASCO-CAP guidelines 2013)
3. Patient must have at least one measurable brain lesion (defined as any lesion ≥ 5mm cm in the longest dimension), on T1 weighted, gadolinium enhanced MRI. Patients may have had surgical excisions of brain metastases provided at least one lesions meets the following criteria:

   * Patients with brain metastases previously untreated with any intra-cranial radiation (i.e. no whole brain radiation therapy [WBRT]/partial brain radiation or stereotactic radiosurgery [SRS]) must have at least one intra-cranial tumor lesion that is ≥ 5mm.
   * Patients with brain metastases previously untreated with any intracranial radiation (i.e., no whole brain radiation therapy [WBRT]/partial brain radiation or stereotactic radiosurgery [SRS]) must have at least one intracranial tumor lesion that is ≥ 5mm.
   * Patients with brain metastases previously treated with WBRT/partial brain radiation only must have at least one intracranial tumor lesion ≥ 5mm and must have evidence of intracranial progressive disease
   * Patients previously treated with WBRT/partial brain radiation and SRS must have at least one intracranial tumor lesion ≥ 5mm that was not treated with SRS and must have intracranial disease.
   * Patients previously treated with SRS must either demonstrate disease progression ≥ 12 weeks after completing SRS with a lesion measuring ≥ 5mm or must have at least one intracranial tumor lesion ≥ 5mm that was not treated with SRS.
4. Patients who have received WBRT/partial brain radiation for intra-cranial metastases are eligible if treatment was completed ≥28 days prior to the first dose of study drug.
5. Estrogen receptor (ER) and progesterone receptor (PR) status in the primary or most recent tumor assessment must be known or pending at the time of study registration. Patient's ER/PR status (i.e., positive or negative) does not influence enrollment but is a requirement.
6. Patient must have received prior treatment with HER2-directed therapy such as trastuzumab, either in the adjuvant or metastatic setting.
7. Prior treatment with lapatinib in the (neo)adjuvant and metastatic setting.
8. Patients without prior chemotherapy for MBC are eligible provided the patients relapsed during adjuvant therapy with trastuzumab or ≤6 months following completion of adjuvant therapy. Otherwise, there is no specific minimum or maximum number of previous chemotherapy regimens for MBC.
9. Patients must have completed cytotoxic chemotherapy ≥21 days (for an every 3-week regimen) or ≥14 days (for an every 2-week or weekly regimen) and have recovered from or come to a new chronic or stable baseline from all treatment-related toxicities in order to be eligible for study treatment.

   * Patient must have completed biologic therapy ≥3 weeks or 5-half lives whichever is shorter.
   * Patient must be discontinued from hormonal therapy a minimum of 1 day prior to the first dose of study treatment.
   * Patients receiving palliative radiation to bone, soft tissue or any other disease sites must have completed this ≥1 week prior to the first dose of study treatment.
10. Patients must have recovered (>2 week recovery is mandated) from any acute neurosurgical intervention for metastatic CNS disease (e.g., resection, shunt placement) and must be clinically stable. These patients must have residual measurable CNS lesion(s) following the surgical procedure if this site is to serve as the target lesion.
11. Patients must be neurologically stable, and if receiving steroids, must be on stable or decreasing doses of corticosteroids and/or anticonvulsants for defined as being on stable low doses of corticosteroids ≥ 5 days prior to the first dose of study treatment.
12. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 2.
13. Adequate hematologic, renal, and hepatic function.
14. Adequate coagulation parameters.
15. Other laboratory testing:

    * Serum magnesium ≥ the institutional lower limit of normal (LLN)
    * Serum potassium ≥ the institutional LLN
16. Left-ventricular-ejection fraction (LVEF) of ≥50% by an echocardiogram (ECHO) or by a multiple-gated acquisition (MUGA)
17. Male patients willing to use adequate contraceptive measures.
18. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start of treatment.
19. Life expectancy ≥12 weeks.
20. Ability to swallow oral medications.
21. Willingness and ability to comply with trial and follow-up procedures.
22. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Previous treatment with cabazitaxel.
2. CNS disease requiring immediate neurosurgical intervention (e.g., resection, shunt placement, etc.).
3. Leptomeningeal metastases as the only site of CNS metastases. Patients with parenchymal brain metastases and leptomeningeal metastases are eligible provided they meet all other eligibility criteria.
4. Peripheral neuropathy ≥Grade 2 (CTCAE v4.0).
5. Concurrent treatment with radiation therapy, hormonal therapy, biologic therapy or chemotherapy is not allowed. Low dose corticosteroids (≤30 mg/day prednisone or its equivalent) are allowed.
6. Concurrent treatment with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A that cannot be discontinued or switched to different medication prior to starting study drug.
7. Concurrent use of St. John's wort and grapefruit/grapefruit juice ≤7 days prior to starting study drug is not allowed.
8. Presence of active gastrointestinal (GI) disease or other condition that in the opinion of the investigator will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, or vomiting).
9. Known diagnosis of human immunodeficiency virus (HIV), Hepatitis B (HBV) or Hepatitis C (HCV).
10. Presence of other active cancers, or history of treatment for invasive cancer ≥3 years. Patients with stage I cancer who have received definitive local treatment with curative intent at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e. non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
11. Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

    * Symptomatic congestive heart failure (CHF) of New York Heart Association Class III or IV.
    * QTc > 480 ms on screening ECG (using the Fredericia formula)
    * Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac or vascular stenting in the past 6 months
    * Active (acute or chronic) or uncontrolled severe infections.
    * Active hepatic or biliary disease (except for patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment).
12. Known hypersensitivity to cabazitaxel or other drugs formulated with polysorbate 80.
13. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
14. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Study Chair — SCRI Development Innovations
Locations (4):
- United States (4):
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Background] Cisternino S, Bourasset F, Archimbaud Y, Semiond D, Sanderink G, Scherrmann JM. Nonlinear accumulation in the brain of the new taxoid TXD258 following saturation of P-glycoprotein at the blood-brain barrier in mice and rats. Br J Pharmacol. 2003 Apr;138(7):1367-75. doi: 10.1038/sj.bjp.0705150. PMID 12711638
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Geyer CE, Forster J, Lindquist D, Chan S, Romieu CG, Pienkowski T, Jagiello-Gruszfeld A, Crown J, Chan A, Kaufman B, Skarlos D, Campone M, Davidson N, Berger M, Oliva C, Rubin SD, Stein S, Cameron D. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006 Dec 28;355(26):2733-43. doi: 10.1056/NEJMoa064320. PMID 17192538
- [Background] Lin NU, Winer EP. Brain metastases: the HER2 paradigm. Clin Cancer Res. 2007 Mar 15;13(6):1648-55. doi: 10.1158/1078-0432.CCR-06-2478. PMID 17363517
- [Background] Lin NU, Carey LA, Liu MC, Younger J, Come SE, Ewend M, Harris GJ, Bullitt E, Van den Abbeele AD, Henson JW, Li X, Gelman R, Burstein HJ, Kasparian E, Kirsch DG, Crawford A, Hochberg F, Winer EP. Phase II trial of lapatinib for brain metastases in patients with human epidermal growth factor receptor 2-positive breast cancer. J Clin Oncol. 2008 Apr 20;26(12):1993-9. doi: 10.1200/JCO.2007.12.3588. PMID 18421051
- [Background] Lin NU, Dieras V, Paul D, Lossignol D, Christodoulou C, Stemmler HJ, Roche H, Liu MC, Greil R, Ciruelos E, Loibl S, Gori S, Wardley A, Yardley D, Brufsky A, Blum JL, Rubin SD, Dharan B, Steplewski K, Zembryki D, Oliva C, Roychowdhury D, Paoletti P, Winer EP. Multicenter phase II study of lapatinib in patients with brain metastases from HER2-positive breast cancer. Clin Cancer Res. 2009 Feb 15;15(4):1452-9. doi: 10.1158/1078-0432.CCR-08-1080. PMID 19228746
- [Background] Pivot X, Koralewski P, Hidalgo JL, Chan A, Goncalves A, Schwartsmann G, Assadourian S, Lotz JP. A multicenter phase II study of XRP6258 administered as a 1-h i.v. infusion every 3 weeks in taxane-resistant metastatic breast cancer patients. Ann Oncol. 2008 Sep;19(9):1547-52. doi: 10.1093/annonc/mdn171. Epub 2008 Apr 23. PMID 18436520
- [Background] Villanueva C, Awada A, Campone M, Machiels JP, Besse T, Magherini E, Dubin F, Semiond D, Pivot X. A multicentre dose-escalating study of cabazitaxel (XRP6258) in combination with capecitabine in patients with metastatic breast cancer progressing after anthracycline and taxane treatment: a phase I/II study. Eur J Cancer. 2011 May;47(7):1037-45. doi: 10.1016/j.ejca.2011.01.001. Epub 2011 Feb 19. PMID 21339064
- [Derived] Yardley DA, Hart LL, Ward PJ, Wright GL, Shastry M, Finney L, DeBusk LM, Hainsworth JD. Cabazitaxel Plus Lapatinib as Therapy for HER2+ Metastatic Breast Cancer With Intracranial Metastases: Results of a Dose-finding Study. Clin Breast Cancer. 2018 Oct;18(5):e781-e787. doi: 10.1016/j.clbc.2018.03.004. Epub 2018 Mar 8. PMID 29678476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2014 and July 2015, 11 subjects with HER2-positive metastatic breast cancer and central nervous system (CNS) metastases were enrolled at 4 investigational sites in the U.S. The study was designed to define the optimal dose of study drugs to administer to subjects, then further assess intracranial response.
Groups:
- Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib): Cabazitaxel: 20 mg/m^2, 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
- Dose Level 2 (Level 1 (25 mg/m^2 Cabazitaxel + Lapatinib): Cabazitaxel: 25 mg/m^2, 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
Period: Overall Study
Arm/Group | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) | Dose Level 2 (Level 1 (25 mg/m^2 Cabazitaxel + Lapatinib)
Started | 6 | 5
Completed | 0 | 0
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive Disease | 3 | 2

BASELINE CHARACTERISTICS:
Population: Includes participants that received at least one dose of study treatment.
Groups:
- Dose Level 1 (20 mg/m2 Cabazitaxel + Lapatinib): Cabazitaxel: 20 mg/m2, 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
- Dose Level 2 (Level 1 (25 mg/m2 Cabazitaxel + Lapatinib): Cabazitaxel: 25 mg/m2, 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (20 mg/m2 Cabazitaxel + Lapatinib) | Dose Level 2 (Level 1 (25 mg/m2 Cabazitaxel + Lapatinib) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 58 [46 to 60] | 60 [40 to 69] | 58 [40 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: CNS Objective Response
Description: The number of patients with Complete and Partial Response (CR+PR) of CNS lesions assessed per modified RECIST Criteria for Evaluation of Intracranial Disease. CR=disappearance of all target and non-target lesions; PR=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter AND an absolute decrease of at least 5mm in at least one target lesion.
Time Frame: every 6 weeks thru cycle 8, then every 9 weeks until treatment discontinuation, projected 1 year
Population: Includes all treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib): Cabazitaxel: 25 mg/m^2, 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
Arm/Group | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib)
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose of Cabazitaxel With Lapatinib
Description: The maximum tolerated dose (MTD) of cabazitaxel and lapatinib will be determined as the highest dose at which ≤1 of 6 patients experiences a dose-limiting toxicity (DLT) assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0. A listing of DLTs are reported in the subsequent Primary Outcome Measure.
Time Frame: weekly for 3 weeks
Population: Includes all treated participants, either at Dose Level 1 or Dose Level 2
Measure: Number; unit: mg/m^2 of cabazitaxel + lapatinib
Groups:
- Cabazitaxel and Lapatinib: Cabazitaxel: (at Dose Level 1, 20 mg/m^2 or at Dose Level 2, 25 mg/m^2), 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
Arm/Group | Cabazitaxel and Lapatinib
Number analyzed (Participants) | 11
mg/m^2 of cabazitaxel + lapatinib | NA — The MTD was not reached. Due to DLTs and other observed toxicities, a decision was made to close the study early.

3. Primary Outcome: Number of Participants Who Experience Dose-Limiting Toxicities (DLTs) as a Measure of Safety
Description: During the safety lead-in, a standard 3+3 dose escalation design is used to determine the maximum tolerated dose (MTD) of cabazitaxel with lapatinib. The MTD would be determined by the highest dose at which ≤1 of 6 patients experiences a dose-limiting toxicity (DLT) during 1 cycle (21 days) of therapy. If 2 of 6 patients within a dose level experiences a DLT, that dose level would be defined as exceeding the MTD and the previous dose level would be evaluated. DLTs are assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.
Time Frame: weekly for 3 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Cabazitaxel: 20 mg/m^2: 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
- Dose Level 2: Cabazitaxel 25mg/m^2:: 1-hour IV infusion on Day 1 of each 3 week cycle, Lapatinib: 1000 mg by mouth (PO) once daily
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 5
Participants
  febrile neutropenia | 0 | 1
  neutropenia | 0 | 1
  diarrhea | 0 | 2
  septic shock | 1 | 0

4. Secondary Outcome: CNS Clinical Benefit Response
Description: The number of patients with Complete Response, Partial Response or Stable Disease extending beyond 6 months (CR+PR+SD ≥ 6 months), determined by RECIST v1.1. CR=disappearance of all target and non-target lesions; PR=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter AND an absolute decrease of at least 5mm in at least one target lesion; SD=Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of the longest diameter since the treatment started.
Time Frame: every 6 weeks thru cycle 8, and every 3 cycles thereafter until treatment discontinuation, projected 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib)
Number analyzed (Participants) | 6 | 5
Participants | 2 | 0

5. Secondary Outcome: Extra-Cranial Objective Response
Description: The number of participants having Complete and Partial Responses (CR+PR) of extra-cranial lesions assessed per RECIST v1.1 Criteria. CR=disappearance of all target and non-target lesions; PR=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter AND an absolute decrease of at least 5mm in at least one target lesion.
Time Frame: every 6 weeks for 8 cycles, then every 9 weeks until treatment discontinuation, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib)
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

6. Secondary Outcome: CNS Progression Free Survival
Description: Evaluate the three and six-month CNS progression free survival measured from date of first protocol treatment until tumor progression or death.
Time Frame: every 6 weeks thru cycle 8, then every 9 weeks until treatment discontinuation, projected 1 year
Population: No data was collected for this outcome measure.
Arm/Group | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Every 3 weeks for approximately 6 months
Description: Adverse events (AEs) were collected for all patients who received at least 1 dose of treatment - from date of first treatment through the 30-day end of treatment period. All patients had at least one AE.
Arm/Group | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib)
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) (N=6) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib) (N=5)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 (1)
DEATH (General disorders) | 1 | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (20 mg/m^2 Cabazitaxel + Lapatinib) (N=6) | Dose Level 2 (25 mg/m^2 Cabazitaxel + Lapatinib) (N=5)
DIARRHOEA (Gastrointestinal disorders) | 5 | 4
FATIGUE (General disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0
BALANCE DISORDER (Nervous system disorders) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0
HOT FLUSH (Vascular disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0
NASAL ULCER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1
SEASONAL ALLERGY (Immune system disorders) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 2
DIZZINESS (Nervous system disorders) | 0 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Early termination of study resulted in small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days